CLINICAL TRIAL: NCT02970513
Title: Psychological Evaluation According Colonic Colonization by Escherichia Coli of Patients After Colorectal Surgery
Acronym: MicrobioPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CHU-0288; 2016-A01233-48 (Other: 2016-A01233-48)
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: Escherichia coli; Microbiota; Colorectal cancer; Psychiatric disorders; Personality traits
MeSH Terms: conditions — Colorectal Neoplasms; Escherichia coli Infections; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients operated on for colorectal cancer (Experimental)
  Interventions: Other: Psychiatric evaluation

INTERVENTIONS:
Other: Psychiatric evaluation — The purpose of this study is to determine whether the presence of pathogenic Escherichia coli in colon is associated with psychiatric disorders.

SUMMARY:
The purpose of this study is to determine whether the presence of pathogenic Escherichia coli in colon is associated with psychiatric disorders.

DETAILED DESCRIPTION:
Colonic colonization by pathogenic Escherichia coli was determined when patients were operated on for colorectal cancer.

Several years later, the investigator investigate past and actual psychiatric disorder using the Mini International Neuropsychiatric Interview (MINI). Actual depression and anxiety scores are evaluated with Hamilton scales and personality traits are investigated using Personality Inventory for DSM-5 (PID-5).

Anxiety and depression scores, psychiatric diagnoses (MINI) and personality traits were compared in patients according to Escherichia coli presence/absence.

ELIGIBILITY:
Inclusion Criteria:

* patients operated on for colorectal cancer in the digestive surgery department of Clermont-Ferrand hospital
* patients older than 18 years,
* patients whose Escherichia coli colonization was analyzed after surgery
* patients which are always followed by the digestive surgery department.

Exclusion Criteria:

* Patients with dementia will not be included, according to the MMSE score:
* 22 if no grade
* 23 if study certificate or CAP or college without patent
* 25 if patent or school without the tray
* 26 or more when bin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Hamilton anxiety and depression score comparison | at day 1
  Hamilton anxiety and depression score will be compared between patients with Escherichi coli colonic colonization and patients without Escherichi coli

SECONDARY OUTCOMES:
Psychiatric prevalence comparison | at day 1
  prevalence of each past and actual psychiatric disorder diagnosed by the Mini International Neuropsychiatric Interview (MINI: major depression, dysthymia, suicidal risk, hypomania, mania, panic disorder, agoraphobia, social phobia, specific phobia, obsessive-compulsive disorder, posttraumatic stress disorder, dependence and abuse of alcohol, tobacco- dependence, psychotic disorders and generalized anxiety disorder) will be compared in patients according to colonic colonization by Escherichia coli.
personality traits comparison | at day 1
  personality traits investigated using Personality Inventory for DSM-5 (PID-5) will be compared in patients according colonic colonization by Escherichia coli

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle JALENQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France